CLINICAL TRIAL: NCT01987609
Title: Evaluation of the Effect of Subcutaneous Hyaluronidase Administration on Psoriatic Plaques
Brief Title: Effects of Subcutaneous Hyaluronidase Administration on Psoriatic Plaques
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tissa Hata, MD (Other)
Responsible Party: Sponsor-Investigator, Tissa Hata, MD, Clinical Professor of Medicine, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCSD 131026
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Results first posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2018-12

CONDITIONS: Psoriasis
Keywords: Psoriasis; Dendritic cells; Hyaluronidase; Hylenex
MeSH Terms: conditions — Psoriasis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hylenex (Experimental): Psoriatic plaques in this arm will be injected with Hylenex every week for 4 weeks.
  Interventions: Drug: Hylenex
- Normal Saline (Placebo Comparator): Psoriatic plaques in this arm will be subcutaneously injected with sterile normal saline every week for four weeks
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Hylenex
  Other Names: Hylenex (R) recombinant; hyaluronidase human injection
  Arms: Hylenex
Drug: Normal Saline
  Other Names: Normal Saline, 0.9%
  Arms: Normal Saline

SUMMARY:
Dendritic cells are a key component of the inflammatory response seen in psoriasis. Several current psoriasis therapies have been shown to reduce the number of dendritic cells in patients with psoriasis, leading researchers to believe that therapies specifically targeting dendritic cells may lead to improvement in psoriasis. Research recently conducted in Dr. Gallo's lab at the University of California San Diego has shown that transgenic mice overexpressing the enzyme hyaluronidase have a significant decrease in the number of dendritic cells in the dermal component of their skin compared to wild type mice. If hyaluronidase overexpression in humans also decreases the number of dendritic cells in the dermis, then hyaluronidase therapy may improve the clinical presentation of psoriasis. In order to test this hypothesis, recombinant human hyaluronidase (Hylenex®) will be injected subcutaneously below a psoriatic plaque in human psoriasis patients every week for a total of 4 weeks. Each week the clinical appearance of the plaque will be documented. At the final visit skin biopsies of the treated plaque will be taken to visualize the histology of the plaque and look for changes in expression of different inflammatory markers.

DETAILED DESCRIPTION:
Participation in this study will consist of a total of 5 visits to the UCSD Dermatology Clinic over approximately a one-month period. At the first visit, two psoriatic plaques between 2-cm and 5-cm in diameter to be studied in this trial will be agreed upon by the patient as well as the blinded and unblinded investigators. Preference will be given to plaques on the elbows since the elbow is a common place of psoriatic plaques, and since scarring on the elbows is usually more acceptable than scarring on other parts of the skin since the skin on the elbows is naturally hyperpigmented in most people. For the remainder of the study, all grading and measurements of the psoriatic plaques will be completed by a blinded investigator who is unaware of which plaque is receiving which treatment. An unblinded investigator will complete all other portions of the study visit, including digital photography, injecting the plaques, and completing the biopsies. The subject will also be blinded as to which plaque is being injected with which treatment.

During the first 4 visits, plaques will be injected with 1-mL of Hylenex® or 1-mL of sterile (pharmaceutical grade) normal saline (NS). 1-mL of Hylenex® contains 150 Units of recombinant hyaluronidase. This is the standard dose of the drug that has been approved by the FDA, and therefore this dose is considered to be safe for use in adults. If injected subcutaneously into the center of a psoriatic plaque that is between 2 and 5 centimeters in diameter, this 1-mL dose should be able to diffuse throughout the entire area beneath the plaque. The exact pharmacokinetics of Hylenex® are difficult to study due to its rapid inactivation after intravenous injection. According to the Hylenex® package insert, though, disruptions to the dermal barrier that occur in response to subcutaneous Hylenex® injection persist 24 hours after injection, but this barrier is completely restored after 48 hours. Cutaneous dendritic cells residing in the epidermis are thought to migrate away from the epidermis through either lymphatic or vascular channels after Hylenex® is injected. This process should take a few hours. Since cutaneous dendritic cells are thought to turnover only every several weeks, new dendritic cells should not populate the epidermis before patients receive the next injection of Hylenex®. Since dendritic cell activation initiates the inflammatory cascade thought to result in psoriasis, preventing dendritic cells from being harbored in the epidermis should essentially prevent the inflammatory cascade that results in psoriasis. Therefore, during the month-long period while patients are receiving Hylenex® injections, the inflammatory cascade triggering their psoriasis will potentially be turned off, allowing affected plaques to heal without propagation of further psoriasis. If this is true, there should be differences in the Hylenex®-treated versus the NS-treated plaques both morphologically and histologically upon completion of the final set of biopsies on the Visit 5.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of plaque psoriasis for at least 6 months, with at least 2 psoriatic plaques on different parts of the body that are both between 2-cm and 5-cm in diameter at the time of screening
* Age 18-65 years
* Male subjects who agree to use barrier methods for contraception throughout the course of the trial if their female partners are of child-bearing potential, or female subjects not of child-bearing potential
* Subject agrees to comply with study requirements
* Subject is fluent in English and is able to provide written informed consent

Exclusion Criteria:

* Subjects with severe medical condition(s) that in the view of the investigator prohibits participation in the study
* Subject has Netherton's syndrome or other genodermatoses that result in a defective epidermal barrier
* Subjects who have applied topical medications (prescription or over-the-counter) for the treatment of psoriasis to their body within 7 days of the baseline visit
* Subjects who have taken cyclosporine, methotrexate, immuran, oral retinoids, chemotherapeutic agents, anti-inflammatory biologics (e.g., alefacept, etanercept, etc.), or oral calcineurin inhibitors within 28 days of the baseline visit
* Subjects who are unable to hold their current psoriasis medications for the period of time indicated (at least 7 days for topical medications, at least 28 days for oral or injectable medications) without significant worsening of their psoriasis
* Immunocompromised subjects (e.g., lymphoma, HIV/AIDS, Wiskott-Aldrich Syndrome), or subjects with a history of malignant disease (excluding non-melanoma skin cancer) as determined by the participant's medical history.
* Subjects receiving phototherapy (e.g., ultraviolet light B [UVB], psoralen plus ultraviolet light A [PUVA]) within 28 days of the baseline visit
* Subjects with a history of psychiatric disease or history of alcohol or drug abuse that would interfere with the ability to comply with the study protocol
* Subjects with significant concurrent medical condition(s) at screening that in the view of the investigator prohibits participation in the study (e.g., severe concurrent allergic disease, condition associated with malignancy, and condition associated with immunosuppression)
* Subjects who have used any systemic antibiotics within 28 days of the baseline visit
* Subjects with an active bacterial, viral or fungal skin infection (excluding nail fungus)
* Subjects currently receiving lithium or have received lithium within the last 4 weeks.
* Ongoing participation in an investigational drug trial
* Subjects with diabetes requiring medication
* Presence of psoriasis with exfoliative erythroderma or presence of guttate psoriasis, primary palmoplantar psoriasis, or pustular psoriasis
* Hypersensitivity to hyaluronidase or any other ingredient in the formulation of hyaluronidase, as well as subjects with an allergy or hypersensitivity to lidocaine
* Subjects taking furosemide, benzodiazepines, phenytoin, salicylates, cortisone, antihistamines or estrogens

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tissa Hata, MD, Principal Investigator — UCSD Division of Dermatology
Locations (1):
- UCSD Division of Dermatology, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: arms
Groups:
- All Study Participants: Psoriatic plaques in one arm of each study participant will be injected with Hylenex every week for 4 weeks.
  Psoriatic plaques on the opposite arm of each study participant will be injected with sterile normal saline every week for 4 weeks.
Period: Overall Study
Arm/Group | All Study Participants
Started | 7; 14 arms (one arm on one patient)
Hylenex Injected in Arm | 6; 6 arms
Normal Saline Injected in Arm | 6; 6 arms
Completed | 6; 12 arms
Not Completed | 1; 2 arms
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: each subject received both treatment and placebo on different arms
Groups:
- All Participants: Each participant had 1 arm randomized to receive Hylenex, and the other hand randomized to receive Normal Saline.
Arm/Group | All Participants
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 7
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Psoriasis Area Severity Index
Description: The Psoriasis Area Severity Index (PASI) of the psoriatic plaques of interest will be measured and compared to baseline values. The PASI is the most widely used tool for the measurement of severity of psoriasis. PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease).
Time Frame: 4 weeks
Measure: Median (Standard Deviation); unit: score on a scale
Units Other Than Participants: arms
Groups:
- Hylenex: Psoriatic plaques in this arm will be injected with Hylenex every week for 4 weeks.
  Hylenex
- Normal Saline: Psoriatic plaques in this arm will be subcutaneously injected with sterile normal saline every week for four weeks
  Normal Saline
Arm/Group | Hylenex | Normal Saline
Number analyzed (Participants) | 7 | 7
Number analyzed (arms) | 7 | 7
score on a scale | 5.5 (2.3) | 5.0 (1.5)

2. Secondary Outcome: Plaque Area
Description: A ruler/measuring tape will be used to measure the area of the subject's psoriatic plaques of interest.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: centimeter^2
Units Other Than Participants: arms
Groups:
- Hylenex: Psoriatic plaques in this arm of each study participant will be injected with Hylenex every week for 4 weeks.
  Hylenex
Arm/Group | Hylenex | Normal Saline
Number analyzed (Participants) | 7 | 7
Number analyzed (arms) | 7 | 7
centimeter^2 | 12.2 (8) | 9.6 (5)

3. Secondary Outcome: Plaque Area
Description: A ruler/measuring tape will be used to measure the area of the subject's psoriatic plaques of interest.
Time Frame: 2 weeks
Measure: Median (Standard Deviation); unit: centimeter^2
Units Other Than Participants: Arms
Arm/Group | Hylenex | Normal Saline
Number analyzed (Participants) | 6 | 6
Number analyzed (Arms) | 6 | 6
centimeter^2 | 9.3 (1.6) | 6.1 (10.8)

4. Secondary Outcome: Plaque Area
Description: A ruler/measuring tape will be used to measure the area of the subject's psoriatic plaques of interest.
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: centimeter^2
Arm/Group | Hylenex | Normal Saline
Number analyzed (Participants) | 6 | 6
centimeter^2 | 13.3 (11.02) | 10.6 (11.35)

5. Secondary Outcome: Plaque Area
Description: A ruler/measuring tape will be used to measure the area of the subject's psoriatic plaques of interest.
Time Frame: 1 weeks
Measure: Mean (Standard Deviation); unit: centimeter^2
Arm/Group | Hylenex | Normal Saline
Number analyzed (Participants) | 7 | 7
centimeter^2 | 11.5 (12.4) | 10.4 (12.5)

6. Secondary Outcome: Physician Global Assessment (PGA)
Description: The Physician Global Assessment (PGA) of the psoriatic plaques of interest will be measured and compared to baseline values on a 0-5 scale where 0 is no evidence of erythema, induration, or scaling, and 5 is severe evidence of these symptoms.
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: psoriatic plaque
Groups:
- Psoriatic Plaques Injected With Hylenex: PGA score of psoriatic plaques on the arm of each study participant that is injected with Hylenex once a week for 4 weeks, at 3 weeks
- Psoriatic Plaques Injected With Normal Saline: PGA score of psoriatic plaques on the arm of each study participant that is injected with normal saline once a week for 4 weeks, at 3 weeks.
Arm/Group | Psoriatic Plaques Injected With Hylenex | Psoriatic Plaques Injected With Normal Saline
Number analyzed (Participants) | 6 | 6
Number analyzed (psoriatic plaque) | 6 | 6
units on a scale | 2.1 (0.9) | 2.2 (0.9)

7. Secondary Outcome: Physician Global Assessment (PGA)
Description: as for outcome 6
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: plaques
Groups:
- Psoriatic Plaques Injected With Hylenex: PGA score of psoriatic plaques on the arm of each study participant that is injected with Hylenex once a week for 4 weeks, at 2 weeks.
- Psoriatic Plaques Injected With Normal Saline: PGA score of psoriatic plaques on the arm of each study participant that is injected with normal saline once a week for 4 weeks, at 2 weeks.
Arm/Group | Psoriatic Plaques Injected With Hylenex | Psoriatic Plaques Injected With Normal Saline
Number analyzed (Participants) | 6 | 6
Number analyzed (plaques) | 6 | 6
units on a scale | 2.1 (1.1) | 2.2 (0.8)

8. Secondary Outcome: Physician Global Assessment (PGA)
Description: as for outcome 6
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: psoriatic plaque
Groups:
- Psoriatic Plaques Injected With Hylenex: PGA score of psoriatic plaques on the arm of each study participant that is injected with Hylenex once a week for 4 weeks, at 1 week.
- Psoriatic Plaques Injected With Normal Saline: PGA score of psoriatic plaques on the arm of each study participant that is injected with normal saline once a week for 4 weeks, at 1 week.
Arm/Group | Psoriatic Plaques Injected With Hylenex | Psoriatic Plaques Injected With Normal Saline
Number analyzed (Participants) | 6 | 6
Number analyzed (psoriatic plaque) | 6 | 6
units on a scale | 2.2 (0.9) | 2.354 (1.1)

9. Secondary Outcome: Change in Histologic Appearance of Psoriatic Plaques
Description: The histologic appearance of a skin biopsy taken from each of the plaques of interest at the end of the study (4 weeks) will be compared to biopsies taken at baseline. The most important feature to be observed is the number of dendritic cells in the different biopsy specimens.
Time Frame: baseline and 4 weeks
Population: Visual data was collected on CD123 staining of dendritic cells in two subjects. Data on the number of dendritic cells were not collected. Further histology/staining was not done given no significant difference was observed in primary endpoint of clinical improvement at interim analysis.
Groups:
- All Participants: Histologic analysis was not done given that no significant difference was observed in primary endpoint of clinical improvement at interim analysis.
Arm/Group | All Participants
Number analyzed (Participants) | 0

10. Secondary Outcome: Change in Tumor Necrosis Factor Alpha (TNFα) Expression
Description: RT-PCR techniques will be used to determine expression levels of the inflammatory cytokine TNFα in all skin biopsies. The expression levels of this cytokine in skin biopsies at week 4 will be compared to the expression levels at baseline.
Time Frame: 4 weeks
Population: Data not collected
Arm/Group | Hylenex | Normal Saline
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change in Interferon Alpha (IFNα) Expression
Description: RT-PCR techniques will be used to determine expression levels of the inflammatory cytokine IFNα in all skin biopsies. The expression levels of this cytokine in skin biopsies at week 4 will be compared to the expression levels at baseline.
Time Frame: 4 weeks
Population: Data not collected.
Arm/Group | Hylenex | Normal Saline
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change in Toll-like Receptor 7 (TLR-7) Expression
Description: RT-PCR techniques will be used to determine expression levels of the TLR-7 in all skin biopsies. The expression levels of this receptor in skin biopsies at week 4 will be compared to the expression levels at baseline.
Time Frame: 4 weeks
Population: Data not collected.
Arm/Group | Hylenex | Normal Saline
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change in Toll-like Receptor 8 (TLR-8) Expression
Description: RT-PCR techniques will be used to determine expression levels of the TLR-8 in all skin biopsies. The expression levels of this receptor in skin biopsies at week 4 will be compared to the expression levels at baseline.
Time Frame: 4 weeks
Population: Data not collected
Arm/Group | Hylenex | Normal Saline
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change in Toll-like Receptor 9 (TLR-9) Expression
Description: RT-PCR techniques will be used to determine expression levels of the TLR-9 in all skin biopsies. The expression levels of this receptor in skin biopsies at week 4 will be compared to the expression levels at baseline.
Time Frame: 4 weeks
Population: Data not collected.
Arm/Group | Hylenex | Normal Saline
Number analyzed (Participants) | 0 | 0

15. Other Pre Specified Outcome: Adverse Events
Description: Any adverse events that subjects have during the course of the study will be recorded at each visit.
Time Frame: 1 week
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Adverse Events
Description: Any adverse events that subjects have during the course of the study will be recorded at each visit.
Time Frame: 2 weeks
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Adverse Events
Description: Any adverse events that subjects have during the course of the study will be recorded at each visit.
Time Frame: 3 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Hylenex | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 1/7 | 1/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hylenex (N=7) | Normal Saline (N=7)
Medication Withdrawal Rebound Flare (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — One subject (subject 5) was terminated early from the study by the investigator due to a rebound flare of psoriasis from medication withdrawal

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT01987609/Prot_SAP_000.pdf